CLINICAL TRIAL: NCT06753552
Title: Combined Effect of Underwater Ultrasound and Custom-made Foot Orthotics in Patients With Rheumatoid Arthritis: A Randomised Controlled Trial
Brief Title: Combined Effect of Underwater Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Researcher, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEU-FTR2
Record Dates: First submitted 2024-12-19; First posted 2024-12-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis of Ankle; Ultrasound Therapy; Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Underwater US+CFO (Experimental)
  Interventions: Other: Underwater US; Device: CFO
- Underwater US (Active Comparator)
  Interventions: Other: Underwater US
- Control (No Intervention)

INTERVENTIONS:
Other: Underwater US — 7 min per session with an intensity of 0.9 W/cm2 for 20 sessions
  Arms: Underwater US; Underwater US+CFO
Device: CFO — Custom made orthotics
  Arms: Underwater US+CFO

SUMMARY:
This randomised controlled trial aims to investigate the effects of underwater ultrasound therapy and customised foot insoles in RA patients. The study evaluates the effects of the combined use of these two methods on pain, functional status and quality of life. The research aims to contribute to current treatment approaches and to demonstrate the effectiveness of innovative methods to improve the quality of life of RA patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that can cause pain, swelling, limitation of movement and deformities in the joints (Cabrera-Sánchez et al. 2024)(Cabrera-Sánchez et al. 2024). Foot and ankle involvement is quite common in RA patients and this may adversely affect the daily living activities of patients. In addition to pharmacological approaches, physical therapy methods and the use of biomechanical supports are also important in the treatment of RA.

Ultrasound is a physical therapy method used to reduce pain and inflammation and accelerate tissue healing (Király et al. 2021). Underwater ultrasound applications may be more effective in superficial areas and may reduce the risk of damage to sensitive tissues around the joint. On the other hand, customised foot insoles (orthotics) are frequently used to correct foot deformities, eliminate biomechanical imbalances and reduce pain (Gaino et al. 2021).

This randomised controlled trial aims to examine the effects of underwater ultrasound therapy and customised foot insoles in RA patients. The study evaluates the effects of the combined use of these two methods on pain, functional status and quality of life. The research aims to contribute to current treatment approaches and to demonstrate the effectiveness of innovative methods to improve the quality of life of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* - ACR/EULAR 2010 diagnostic criteria with foot involvement and having a disease duration of less than two years were enrolled in the study over a period of three months.
* with foot involvement diagnosed by a rheumatologist.

Exclusion Criteria:

* - Degenerative diseases and anatomical abnormalities were excluded
* if they presented in an acute symptomatic flare or they needed to use walking assistance
* neurological problems, malignant process, cognitive deterioration, pregnancy, previous foot surgery and the presence of a foot wound

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
DAS-28 | 4 weeks
  Measures disease activity by evaluating 28 joints for swelling and tenderness.
Manchester-Oxford Foot Questionnaire (MOXFQ) | 2 weeks
Health Assessment Questionnaire [HAQ] | 2 weeks
Berg Balance Test | 4 weeks
  Useful for the measurement of the risk of falls and for demonstrating the progress patients in exercise programs oriented to the improve of balance for falls prevention.

SECONDARY OUTCOMES:
Ankle Girth Measurement | 4 weeeks
  https://orthofixar.com/special-test/ankle-girth-measurement/
Timed Up and Go Test | 4 weeks
  Measures overall mobility and fall risk.
Quebec User Evaluation of Satisfaction: | 4 weeks
  Satisfaction of the custom made insoles

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Ahi Evran, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
via e-mail perhaps